CLINICAL TRIAL: NCT06718088
Title: Risk Factors Associated With The Progression Of Adenomyosis
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PROADENO
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Adenomyosis
Keywords: adenomyosis; risk factors; transvaginal ultrasound
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adenomyosis is a gynaecological disorder with a high prevalence in women of childbearing age and is characterised by the presence of endometrial glands and stroma within the myometrium, associated or not with hypertrophy and hyperplasia of the surrounding myometrium. Adenomyosis may cause pelvic pain and/or abnormal uterine bleeding.

Transvaginal ultrasound (TVUS) is considered the main non-invasive diagnostic modality for the diagnosis of adenomyosis.

Although adenomyosis is a very common condition among patients of childbearing age, its natural course is still debated. Some studies have evaluated the role of hormonal treatments (systemic or local oestrogen or progestin-based) on adenomyosis, which have been effective in controlling symptoms such as pelvic pain and abnormal uterine bleeding. Despite all this, no evidence is available on the progression of adenomyosis and the factors that may influence its progression over time. The aim of this study is therefore to assess the progression of adenomyosis and associated risk factors using transvaginal ultrasound.

DETAILED DESCRIPTION:
Adenomyosis is a gynaecological disorder with a high prevalence in women of childbearing age and is characterised by the presence of endometrial glands and stroma within the myometrium, associated or not with hypertrophy and hyperplasia of the surrounding myometrium. Adenomyosis may cause pelvic pain and/or abnormal uterine bleeding.

Transvaginal ultrasound is considered the main non-invasive diagnostic modality for the diagnosis of adenomyosis.

The goal of formulating a recognised and unified terminology for the description of ultrasound criteria for the diagnosis of adenomyosis was achieved by the Morphological Uterus Sonographic Assessment (MUSA) consensus.

The MUSA consensus consists of a list of ultrasound features associated with adenomyosis, namely:

* globular uterus: uterus with a more spherical conformation and more slender bottom than normal. The definition of a 'globular uterus' is currently subjective and there are no quantitative uterine biometric parameters available to differentiate a uterus with adenomyosis from a uterus not affected by the disease (normal or fibromatous uterus).
* asymmetric thickening of the uterine walls;
* inhomogeneous eco-structure due to the presence of multiple hyperechogenic striae intermixed with hypoechogenic striae (thin shadow cones) giving the typical ultrasound appearance described as 'rain in the forest' or 'fan-shaped shadowing';
* cystic spaces or non-vascularised intra-myometrial anecogenic lacunae, often surrounded by a hyper-echogenic halo, caused by glandular ectasia;
* hyperechogenic islands deepening in the myometrium, expression of the presence of islands of ectopic endometrial tissue;
* subendometrial lines and spicules;
* intralesional and irregular vascularisation of the myometrium (vessels penetrate in a rectilinear within adenomyomas or foci of adenomyosis);
* poor definition of the endometrium/myometrium junction (JZ);
* thickening, irregularities and interruptions of the JZ.

To these ultrasound features summarised by the MUSA consensus, the literature adds two that are considered equally typical of the pathology:

* uterine pain on pressure of the ultrasound probe;
* the 'question mark sign', i.e. a pathological angle at the uterine fundus, an expression of uterine anatomical distortion.

Previous studies on the occurrence of adenomyosis have been limited to women undergoing hysterectomy, probably overestimating its prevalence compared to the general population. Recent studies, on the other hand, have begun to investigate the morphological features of adenomyosis using TVUS, an inexpensive and widely available method, to determine its prevalence and the factors that may influence its onset. They defined a prevalence of the condition as 20.9% among women attending a gynaecological outpatient setting.

Although adenomyosis is a very common condition among patients of childbearing age, its natural evolution is still debated. Some studies have evaluated the role of hormonal treatments (systemic or local oestrogen or progestin-based) on adenomyosis, which have been effective in controlling symptoms such as pelvic pain and abnormal uterine bleeding. Despite all this, no evidence is available regarding the progression of adenomyosis and the factors that may influence its progression over time. The aim of this study is therefore to assess the progression of adenomyosis and associated risk factors using transvaginal ultrasound.

The study is prospective and retrospective observational.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 55 years;
* Presence of at least two direct and indirect signs according to the MUSA classification
* Obtaining informed consent

Exclusion Criteria:

* Patients undergoing hysterectomy;
* Virgo patients;
* Patients reporting intolerance to transvaginal ultrasound;
* Gynaecological oncology;
* Recent pregnancy or childbirth (within 6 months)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with ultrasound diagnosis of adenomyosis who were referred to the ultrasound outpatient clinics for routine check-ups or pre-operative visits, as per their regular care routine.
  The retrospective arm of the study will enrol patients who have been admitted to our outpatient clinics since 1 January 2018. The ultrasound diagnosis of adenomyosis will be made if at least 2 ultrasound signs compatible with adenomyosis are present according to the modified MUSA consensus.
  Women included in the study will be offered ultrasound follow-up at 6, 12, 24, 36, 48 months after the first outpatient visit with a diagnosis of adenomyosis. Subsequently, patients will be divided into three groups according to evidence of progression, stability and regression of the adenomyotic picture at follow-up
Sampling Method: Non-Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression of adenomyosis | At 12, 24, 36 and 48 months
  Risk of progression of adenomyosis and the risk factors associated with progression in patients with ultrasound diagnosis of adenomyosis

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Casadio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy